CLINICAL TRIAL: NCT06693804
Title: Quality Improvement Initiative: Using Digital Ophthalmoscope and Otoscope Visual Arts Observation Training to Improve Family Medicine Residency Training
Brief Title: Ophthalmoscope and Otoscope Training in Family Medicine Residency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Wiedemer, MD, Associate Professor, Program Director of Penn State Health Family and Community Medicine Residency at Mount Nittany Medical Center, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00020873
Record Dates: First submitted 2024-11-10; First posted 2024-11-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Resident Education; Digital Technology
Keywords: otoscope; ophthalmoscope; visual arts; resident; device; instrument; eye exam; ear exam; family medicine; education
MeSH Terms: interventions — Ophthalmoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Welch Allyn PanOptic iExaminer Digital Imaging Kit (Experimental): Novel digital instrument to visualize eyes and ears in clinical practice
  Interventions: Other: Digital Otoscope and Ophthalmoscope
- Conventional non-digital instrument used in current clinical training and standard practice (Active Comparator): Standard practice
  Interventions: Other: Conventional otoscope and ophthalmoscope

INTERVENTIONS:
Other: Digital Otoscope and Ophthalmoscope — The otoscope and ophthalmoscope will be used by residents to examine the eyes and ears under illumination and magnification during physical examinations.
  Arms: Welch Allyn PanOptic iExaminer Digital Imaging Kit
Other: Conventional otoscope and ophthalmoscope — The otoscope and ophthalmoscope will be used by residents to examine the eyes and ears under illumination during physical examinations.
  Arms: Conventional non-digital instrument used in current clinical training and standard practice

SUMMARY:
The purpose of the study is to evaluate the effectiveness of Welch Allyn PanOptic Plus Ophthalmoscope with smartphone adaptor, and assess residents' opinions on acceptability and usability of the device and curriculum vs the conventional non-digital device used in current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Resident in Penn States Family and Community Medicine Department

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Resident Confidence Survey (Pre) | 0 months
  Survey will measure Resident's confidence. Survey will consist of 10 questions based on a Likert scale where a value of 1=not at all confident and 5=very confident. A score of 10 would indicate no confidence and a score of 50 would indicate complete confidence.
Resident Knowledge Survey (Post) | 3 months
  Survey will measure Resident's knowledge. Survey will consist of 12 questions based on a Likert scale where a value of 1=not at all confident and 5=very confident. A score of 12 would indicate absence of knowledge and a score of 60 would indicate complete knowledge.
Visual Identification of Images (Pre) | 0 months
  Residents will be shown 34 images of the eye and ear which they will need to correctly identify. Correct identification of 0 images = lowest score. Correct identification of 34 images = highest score.
Visual Identification of Images (Post) | 3 months
  Residents will be shown 34 images of the eye and ear which they will need to correctly identify. Correct identification of 0 images = lowest score. Correct identification of 34 images = highest score.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wiedemer, MD, Principal Investigator — The Pennsylvania State University, College of Medicine, Family and Community Medicine Department
Locations (2):
- United States (2):
  - Penn State Milton S. Hershey Medical Center, Harrisburg, Pennsylvania
  - Penn State Health St. Joseph Medical Center, Reading, Pennsylvania